CLINICAL TRIAL: NCT01623531
Title: The Use of Fibrinogen Concentrate in High-Risk Cardiac Surgery. A Prospective, Double-blinded, Randomized, Controlled Study
Brief Title: Prospective Double Blinded Randomized Control Study of the Use of Fibrinogen in High-Risk Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Myron Kwapisz, MD, MD, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fibrinogenstudy0911
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Complication During Procedure
Keywords: Fibrinogen; cardiac surgery; high risk; cardiopulmonary bypass; bleeding; blood transfusion
MeSH Terms: conditions — Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RiaSTAP (Active Comparator): Intravenous fibrinogen(RiaSTAP) will be administered according to FIBTEM based calculation formula
  Interventions: Drug: Fibrinogen
- Intravenous saline (Placebo Comparator): Intravenous saline (placebo) will be calculated according to FIBTEM based calculation formula
  Interventions: Drug: Fibrinogen

INTERVENTIONS:
Drug: Fibrinogen — Intravenous concentrated fibrinogen will be infused according to a hemostatic algorithm based on ROTEM (FIBTEM)
  Other Names: RiaSTAP or Haemocomplettan P

SUMMARY:
The aim of the study is to show that first line treatment with concentrated fibrinogen has superiority over the conventional therapy with fresh frozen plasma (FFP), platelets, and cryoprecipitate in perioperative management of bleeding after complex cardiac surgery.

DETAILED DESCRIPTION:
All patients will be recruited from the Queen Elizabeth II (QEII) Health Sciences Center, Halifax, Nova Scotia, which is the sole tertiary cardiac surgical referral center in Nova Scotia that performs approximately 1000 open heart surgical procedures yearly, including more than 700 isolated coronary artery bypass graft (CABG) procedures.

Inclusion criteria: All patients who are scheduled for elective complex cardiac surgical procedures including, double procedures (aortic valve replacement+coronary artery bypass graft , mitral valve replacement+coronary artery bypass graft , aortic valve replacement+mitral valve replacement), redo-sternotomies, and aortic root repair +/-aortic valve replacement.

Exclusion criteria: Any known congenital or preexisting bleeding disorder, preexisting clinically significant abnormal fibrinogen level, severe liver disease (alanine aminotransferase or aspartate aminotransferase > 150 U/l), inability of providing informed consent, emergency surgery, pregnancy or nursing, age under 18 years, intake of anti-platelet drugs within the last 2- 5 days before surgery (low dose aspirin is allowed) allergy to concentrated fibrinogen or other components in the product, anemia (Hb < 110), diagnosed deep venous thrombosis, pulmonary embolism, acute stroke or acute myocardial infarction.

The primary outcome: Cumulative perioperative amount (number of units and total volume) of blood components used between the start of surgery and 24 hours after administration of the study drug or placebo. 'Blood Components' are defined as all fresh components of blood (RBCs, plasma, platelets, and Cryo).

The secondary outcomes: Fibrinogen levels, hematocrit, prothrombin time (PT), partial prothrombin time (PTT), INR, platelet count, Hemoglobin (Hb), Thromboelastometry (ROTEM®, clotting time (CT), clot formation time (CFT), Angle, maximum clot firmness (MCF), Cardiovascular intensive care unit (CVICU-stay), Hospital-stay, In-Hospital Mortality, Hemoglobin, adverse events (anaphylaxis, stroke, myocardial infarction, pulmonary embolism, and deep vein thromboembolism) and usage of factor VII concentrate and human prothrombin complex (factors II, VII,IX, X), total avoidance of transfusion after cardiopulmonary bypass (CPB) 24h after administration of study drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

All patients who are scheduled for elective complex cardiac surgical procedures including

* double procedures (aortic valve replacement (AVR)+CABG, mitral valve repair/replacement (MVR)+CABG, AVR+MVR)
* Redo-sternotomies
* Aortic root repair +/- AVR

Exclusion Criteria:

* Any known congenital or pre-existing bleeding disorder
* pre-existing clinically significant abnormal fibrinogen level (normal: 2.5-4.79g/l)
* severe liver disease (alanine aminotransferase or aspartate aminotransferase > 150 U/l)
* inability to provide informed consent
* emergency surgery
* pregnancy or nursing
* age under 18 years
* intake of anti-platelet drugs within2- 5 days preoperatively (low dose ASA is allowed)
* allergy to concentrated fibrinogen or other components in the product
* anemia (Hgb < 110)
* diagnosed deep vein thrombosis (DVT)
* pulmonary embolism
* acute stroke
* acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-02; Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Kwapisz, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- CapitalDHACanada, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Kwapisz MM, Kent B, DiQuinzio C, LeGare JF, Garnett S, Swyer W, Whynot S, Mingo H, Scheffler M. The prophylactic use of fibrinogen concentrate in high-risk cardiac surgery. Acta Anaesthesiol Scand. 2020 May;64(5):602-612. doi: 10.1111/aas.13540. Epub 2020 Jan 17. PMID 31889306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigation included 62 patients (>18 years old) for elective, high-risk cardiac surgery (double procedures (aortic valve replacement (AVR)+coronary artery bypass grafting (CABG), mitral valve repair/replacement (MVR)+CABG, AVR+MVR), redo-sternotomies, and aortic root repair±AVR) with a pre-operative fibrinogen level of ≤3.8 g/L.
Groups:
- Intravenous Saline: Intravenous saline (placebo) will be calculated according to FIBTEM based calculation formula
  Placebo: Intravenous saline will be administered with the same volume as study drug
Period: Overall Study
Arm/Group | RiaSTAP | Intravenous Saline
Started | 31 | 31
Completed | 27 | 29
Not Completed | 4 | 2
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Missing data at primary outcome time poi | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intravenous Saline: Intravenous saline (placebo) will be calculated according to FIBTEM based calculation formula
  Placebo: Intravenous saline will be infused with the same volume of the study drug.
- Total: Total of all reporting groups
Arm/Group | RiaSTAP | Intravenous Saline | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (18) | 65 (11) | 62 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 23 | 27 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 28 | 30 | 58
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (4.14) | 29 (4.03) | 28.9 (4)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Transfusion Units
Description: Including packed red cells, frozen plasma, platelets, cryoprecipitates
Time Frame: 24 hours after administration of study drug
Measure: Median (Inter-Quartile Range); unit: Transfusion Units
Groups:
- Intravenous Saline: Intravenous saline (placebo) will be calculated according to FIBTEM based calculation formula
  Placebo: Intravenous placebo will be infused with the same volume as the study drug.
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
Transfusion Units | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; Normality among study outcomes was investigated with Shapiro-Wilk tests, histograms, boxplots, and graphing of residuals, revealing that the data were not normally distributed, and primary outcomes were zero inflated. Therefore, we used non-parametric Mann-Whitney U-tests with a 2-sided type I error rate of 5%. We tested the null hypothesis of no difference in primary and secondary outcomes between groups 24 hours after infusion of the study drug; Test type: Superiority; p = .908, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 386, Standard Error of Mean 47.50 — The distributions of cumulative transfusion units did not differ significantly between patients receiving either RiaSTAP (median = 0, IQR = 0-1) or Placebo (median = 0, IQR = 0.1), U = 386, SE = 47.60, p = .908

2. Secondary Outcome: Fibrinogen Plasma Concentration (g/L)
Time Frame: 24h after infusion of study drug
Population: Six patients had missing data in the fibrinogen group (RiaStap) at 24h after infusion of study drug. Six patients had missing data in the placebo group at 24h after infusion of study drug.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 22 | 24
g/L | 4.65 (0.94) | 4.15 (0.68)
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; We tested the null hypothesis of no difference in primary and secondary outcomes between groups 24 hours after infusion of the study drug. Normality among study outcomes was investigated with Shapiro-Wilk tests, histograms, boxplots, and graphing of residuals. For normally distributed data unequal variance t tests were used; Test type: Superiority; p = .047, t-test, 2 sided; Unequal variances assumed; Mean Difference (Net) = -.498, Standard Error of Mean .239 — Unequal variances T-test comparing placebo to RiaSTAP

3. Secondary Outcome: Hematocrit (%)
Time Frame: 24h after infusion of study drug
Population: Four patients in the fibrinogen group (RiaStap) had missing data at 24h after infusion of study drug. Two patients in the placebo group had missing data at 24h after infusion of study drug.
Measure: Mean (Standard Deviation); unit: Hematocrit percent
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 24 | 28
Hematocrit percent | 0.29 (0.04) | 0.28 (0.05)
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .729, t-test, 2 sided; Unequal variances assumed; Mean Difference (Net) = -.004, Standard Error of Mean .0116 — Unequal variances T-test comparing placebo to RiaSTAP

4. Secondary Outcome: Hemoglobin Concentration (g/L)
Time Frame: 24h after infusion of study drug
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 24 | 28
g/L | 95 (11.9) | 95 (14.8)
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .93, t-test, 2 sided; Unequal variances assumed; Mean Difference (Net) = -.321, Standard Error of Mean 3.699 — Unequal variances T-test comparing placebo to RiaSTAP

5. Secondary Outcome: Platelet Count (10^3/μL)
Time Frame: 24h after infusion of study drug
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells*10^3/μL
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 24 | 28
cells*10^3/μL | 129 (31.4) | 117 (29.3)
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; Test type: Superiority; p = .169, t-test, 2 sided; Unequal variances assumed; Mean Difference (Net) = -11.821, Standard Error of Mean 8.471 — Unequal variances T-test comparing placebo to RiaSTAP

6. Secondary Outcome: Partial Thromboplastin Time (s)
Time Frame: 24h after infusion of study drug
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 24 | 28
seconds | 31 [27 to 33] | 28.5 [27 to 30]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; Normality among study outcomes was investigated with Shapiro-Wilk tests, histograms, boxplots, and graphing of residuals, revealing that this variable was not normally distributed. Therefore, we used non-parametric Mann-Whitney U-tests with a 2-sided type I error rate of 5%. We tested the null hypothesis of no difference in secondary outcomes between groups 24 hours after infusion of the study drug; Test type: Superiority; p = .035, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 450.5, Standard Error of Mean 54.163

7. Secondary Outcome: International Normalized Ratio
Description: International normalized ratio (INR) is calculated based on the prothrombin time (PT) test results.The PT is usually measured in seconds and is compared to a normal range that reflects PT values in healthy individuals. Because the reagents used to perform the PT test vary from one laboratory to another and even within the same laboratory over time, the normal ranges also will fluctuate. To standardize results across different laboratories in the world, a World Health Organization (WHO) committee developed and recommended the use of the Internationalized Normalized Ratio (INR). The INR is calculated with the ratio of the patient's prothrombin time (PT test) to a normal prothrombin time (control) sample (PT normal): INR=PT test:PT normal. The normal range is from 0.9 to 1.2. The higher the value the more is the patient anticoagulated. This means the patient's blood is thinner with a lower concentration of coagulation factors.
Time Frame: 24h after infusion of study drug
Population: Four patients in the fibrinogen group (RiaStap) had missing data at 24h after infusion of study drug. Three patients in the placebo group had missing data at 24h after infusion of study drug.
Measure: Median (Full Range); unit: Ratio
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 24 | 27
Ratio | 1.2 [1.0 to 1.9] | 1.2 [1.0 to 1.5]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .794, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 337.5, Standard Error of Mean 51.591

8. Secondary Outcome: Prothrombin Time (s)
Description: The prothrombin time (PT) test evaluates how well all of the coagulation factors in the extrinsic and common pathways of the coagulation cascade work together. Included are: factors I (Fibrinogen), II (Prothrombin), V, VII and X.
Time Frame: 24h after infusion of study drug
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 24 | 27
seconds | 13.9 [13 to 15] | 13.8 [13 to 15]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .828, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 335.5, Standard Error of Mean 52.957

9. Secondary Outcome: EXTEM Clotting Time (s)
Description: EXTEM = rotational thrombelastometry (measurement of extrinsic coagulation pathway); clotting time: time from start of the measurement until initiation of clotting (thrombin formation, start of clot polymerisation).
Time Frame: 24h after infusion of study drug
Population: One patient in the fibrinogen group (RiaStap) had missing data at 24h after infusion of study drug. One patient in the placebo group had missing data at 24h after infusion of study drug.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
seconds | 68 [63 to 74] | 68 [62 to 75]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .941, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 396, Standard Error of Mean 60.944

10. Secondary Outcome: EXTEM Maximum Clot Firmness (mm)
Description: EXTEM = rotational thrombelastometry (measurement of extrinsic coagulation pathway); maximum clot firmness: increasing stabilisation of the clot by the polymerised fibrin, platelets as well as factor XIII.
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
mm | 66 [63 to 70] | 64 [61 to 67]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .09, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 494.5, Standard Error of Mean 60.783

11. Secondary Outcome: INTEM Clotting Time (s)
Description: INTEM = rotational thrombelastometry (measurement of intrinsic coagulation pathway); clotting time: time from start of the measurement until initiation of clotting (thrombin formation, start of clot polymerisation).
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
seconds | 161 [146 to 175] | 164 [148 to 167]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .658, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 418.500, Standard Error of Mean 60.93

12. Secondary Outcome: INTEM Maximum Clot Firmness (mm)
Description: INTEM = rotational thrombelastometry (measurement of intrinsic coagulation pathway); maximum clot firmness: increasing stabilisation of the clot by the polymerised fibrin, platelets as well as factor XIII.
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
mm | 64 [63 to 68] | 63 [50 to 66]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .182, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 472.5, Standard Error of Mean 60.727

13. Secondary Outcome: FIBTEM Clotting Time (s)
Description: FIBTEM = rotational thrombelastometry (measurement of functional fibrinogen); clotting time: time from start of the measurement until initiation of clotting (thrombin formation, start of clot polymerisation).
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
seconds | 64 [56 to 67] | 59 [54 to 67]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .549, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 428, Standard Error of Mean 60.919

14. Secondary Outcome: FIBTEM MCF (Maximum Clot Firmness)
Description: Rotational thrombelastometry (measurement of functional fibrinogen). Rotational thrombelastometry (ROTEM) is a point-of-care viscoelastic coagulation test. The device provides four channels for simultaneous assays. With the so called "FIBTEM" assay coagulation is activated by a small amount of tissue thromboplastin (tissue factor) and platelets are blocked with cytochalasin D. The resulting clot is therefore only depending on fibrin formation and fibrin polymerisation. The maximum clot firmness (MCF) is the amplitude in mm on the result graph representing the increasing stabilisation of the clot.
Time Frame: 24 hours after study drug administration
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- Intravenous Saline: Intravenous saline (placebo) will be calculated according to FIBTEM based calculation formula
  Placebo: Intravenous saline will be infused with the same volume as the study drug.
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
mm | 27 [24 to 30] | 23 [22 to 27]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; Normality among study outcomes was investigated with Shapiro-Wilk tests, histograms, boxplots, and graphing of residuals, revealing that the FIBTEM MCF data was not normally distributed. Therefore, we used non-parametric Mann-Whitney U-tests with a 2-sided type I error rate of 5%. We tested the null hypothesis of no difference in secondary outcomes between groups 24 hours after infusion of the study drug; Test type: Superiority; p = .022, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 530.5, Standard Error of Mean 60.816 — The distribution of FIBTEM MCF (maximum clot firmness) was significantly different between RiaSTAP (median = 27 mm, IQR = 24, 30), and placebo (median = 23 mm, IQR = 22, 27) groups, U-test = 530.5, SE = 60.816, p = .022)

15. Secondary Outcome: HEPTEM Clotting Time (s)
Description: HEPTEM = rotational thrombelastometry (measurement of INTEM with heparinase);clotting time: time from start of the measurement until initiation of clotting (thrombin formation, start of clot polymerisation).
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
seconds | 162 [152 to 184] | 162 [149 to 172]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .455, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 437, Standard Error of Mean 60.930

16. Secondary Outcome: HEPTEM Maximum Clot Firmness (mm)
Description: HEPTEM = rotational thrombelastometry (measurement of INTEM with heparinase); maximum clot firmness: increasing stabilisation of the clot by the polymerised fibrin, platelets as well as factor XIII.
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
mm | 62 [58 to 67] | 61 [58 to 63]
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = .5, Wilcoxon (Mann-Whitney); Mann-Whitney U test = 432.5, Standard Error of Mean 60.819

17. Secondary Outcome: Total Avoidance of Transfusions
Description: Total avoidance of any transfusion after cardiopulmonary bypass (CPB) 24h after administration of study drug or placebo.
Time Frame: 24h after infusion of study drug
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
Participants
  Avoided transfusions | 20 | 21
  Had any transfusion | 7 | 8
Statistical Analysis 1: Comparison: RiaSTAP vs Intravenous Saline; Test type: Superiority; p = 1.0, Fisher Exact; Significance (2-sided) using Fisher's Exact Test

18. Other Pre Specified Outcome: Overall Numbers of Patients Receiving Blood Products
Description: Including Packed Red Cells, Fresh Frozen Plasma, Platelets, Cryoprecipitate and coagulation factor concentrates. The study was not sufficiently powered to test differences between this outcome.
Time Frame: 24 hours after administration of study drug
Population: The placebo group had one dropout during the study because of a study protocol violation and one patient with missing data at the primary outcome time point (29pt). The fibrinogen group hat three dropouts during the study because of two study protocol violation, one death and one patient with missing data at the primary outcome time point (27pt).
Measure: Count of Participants; unit: Participants
Arm/Group | RiaSTAP | Intravenous Saline
Number analyzed (Participants) | 27 | 29
Participants | 7 | 8

ADVERSE EVENTS:
Time Frame: All study patients were followed with a phone call interview after 6 weeks, 3, and 6 months post-operatively. All patients were assessed for the following events: angina, re-admission (congestive heart failure [CHF], acute myocardial infarction [AMI], acute coronary syndrome [ACS], and percutaneous coronary intervention [PCI]), incisional wound infection, thromboembolic complications (pulmonary embolism, deep venous thrombosis), repeated cardiac surgery, and cardiac mortality.
Arm/Group | RiaSTAP | Intravenous Saline
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 5/27 | 9/29
Other Adverse Events (participants affected / at risk) | 1/27 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RiaSTAP (N=27) | Intravenous Saline (N=29)
Re-Operation (Surgical and medical procedures) | 1 (1) | 4 (4) — Re-exploration with Re-sternotomy because of acute cardiac tamponade or diffuse or surgical bleeding
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Upper extremity weakness
Postoperative Delirium (Psychiatric disorders) | 2 (2) | 5 (5)
Death (Nervous system disorders) | 1 | 0 — Generalized, diffuse brain edema on postop. day 1 after hemi aortic arch repair
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RiaSTAP (N=27) | Intravenous Saline (N=29)
Incisional wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was limited by a less than expected transfusion rate and the inability to reach the planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT01623531/Prot_SAP_000.pdf